CLINICAL TRIAL: NCT05088486
Title: Preventive and Personalized Medicine (2021-2023)
Brief Title: The Role of Genetic Factors in the Development of Arterial Hypertension in the Kazakh Population
Status: Completed | Type: Observational
Sponsor: Asfendiyarov Kazakh National Medical University (Other)
Responsible Party: Principal Investigator, Ildar Fakhradiyev, Head of the Laboratory of Experimental Medicine, Asfendiyarov Kazakh National Medical University
Other Study IDs: 1193
Record Dates: First submitted 2021-09-25; First posted 2021-10-22 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Arterial Hypertension
Keywords: GWAS
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group:: Patients with arterial hypertension
  Interventions: Genetic: DNA analysis
- Control group: Patients without arterial hypertension
  Interventions: Genetic: DNA analysis

INTERVENTIONS:
Genetic: DNA analysis — GWAS

SUMMARY:
This is a GWAS study that aims to identify possible candidate genes associate to arterial hypertension by exploring single nucleotide polymorphism (SNP) in a group of arterial hypertension, in the Kazakh population. The investigators hypothesize that the careful phenotyping of the subject sand matching with increase the power to find SNP significantly associate with arterial hypertension

DETAILED DESCRIPTION:
A genome-wide association study (GWAS) is an approach used in genetics research to associate specific genetic variations with particular diseases. The method involves scanning the genomes from many different people and looking for genetic markers that can be used to predict the presence of a disease. Once such genetic markers are identified, they can be used to understand how genes contribute to the disease and develop better prevention and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Persons with confirmed arterial hypertension;
* The age of patients is from 18 to 55 years old inclusive;
* Persons of Kazakh nationality, whose paternal and maternal grandparents identify themselves as Kazakhs;
* Persons who are able and willing to provide written informed consent;
* Persons capable and willing to comply with the research protocol;

Exclusion Criteria:

* Persons under 18 and over 55;
* Persons who, in the opinion of the researcher, are mentally or legally incapacitated, which prevents obtaining informed consent;
* Pregnant or lactating women;
* Tuberculosis of any localization in the active phase and in history;
* Severe and decompensated diseases of the liver and kidneys, cardiovascular system;
* Severe and decompensated course of endocrine diseases;
* Autoimmune diseases;
* Systemic diseases;
* Cancer.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: patients with arterial hypertension of Kazakh nationality
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
number of SNPs associated with arterial hypertension | 1 year
  Using GWAS to identify candidate genes associate with arterial hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Raushan Karibayeva, Doctor of medical sciences, Study Director — Deputy head of Gerontology Center of Medical Centre Hospital of the President's Affairs Administration of the Republic of Kazakhstan; Tamara Vochshenkova, MBA, Study Chair — Deputy head of Gerontology Center of Medical Centre Hospital of the President's Affairs Administration of the Republic of Kazakhstan
Locations (1):
- Deputy head of Gerontology Center of Medical Centre Hospital of the President's Affairs Administration of the Republic of Kazakhstan, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided